CLINICAL TRIAL: NCT04051073
Title: Can Continuous Non-invasive Monitoring Improve Stability of Intraoperative Blood Pressure - A Feasibility Study.
Acronym: iSTABILISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: University of Warwick (Other)
Responsible Party: Principal Investigator, William Rook, Academic Clinical Fellow, University of Warwick
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2019003AN
Record Dates: First submitted 2019-07-26; First posted 2019-08-09 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Hip Fractures; Hypotension on Induction; Intraoperative Hypotension; Acute Kidney Injury; Myocardial Ischemia; Wound Infection; Perioperative/Postoperative Complications
MeSH Terms: conditions — Hip Fractures; Acute Kidney Injury; Myocardial Ischemia; Wound Infection; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Before-and-after
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blinded (Sham Comparator): CNAP monitoring applied, but screen and information not visible to treating anaesthetist
  Interventions: Device: Continuous non-invasive blood pressure monitoring
- Unblinded (Active Comparator): CNAP monitoring applied and available in full to the treating anaesthetist
  Interventions: Device: Continuous non-invasive blood pressure monitoring

INTERVENTIONS:
Device: Continuous non-invasive blood pressure monitoring — Continuous non-invasive blood pressure monitoring using CNAP

SUMMARY:
Background During anaesthesia for repair of a broken hip, many patients experience low blood pressure. There have been many studies showing that patients who experience low blood pressure during anaesthesia are at increased risk of sustaining kidney or heart damage, strokes, having a post-operative infection, or dying. During anaesthesia, in most cases blood pressure is monitored using a cuff which inflates on the arm (the 'normal' way blood pressure is measured in a GP practice or hospital ward). This gives a reading each time the cuff goes up and down, every 3-5 minutes typically. There is a less well used way to measure blood pressure, using an additional cuff on the finger which gives a constant, continuous measure of blood pressure. We think that using this monitor, rather than the 'standard' monitor, will mean that low blood pressure is recognised more quickly, therefore treated more quickly, and will lead to patients having less exposure to dangerously low blood pressures. If this is the case, we hope that it will reduce how often patients experience kidney or heart damage, have an infection after surgery, suffer a stroke, and reduce the risk of death.

Methodology To test this, we would need to run a large clinical trial comparing the continuous monitor to the standard monitor. This would be expensive and involve a great deal of work in a large number of hospitals, and so first we wish to determine whether the trial we would like to run is practical, and possible to deliver in the real world. To do this we plan to run the trial first on a small-scale feasibility (pilot) study, where we will recruit 30 patients, half of whom will have the standard monitor, and half of whom will have the continuous monitor. We will see what proportion of the patients who could enter the trial actually do so and complete it, and use it as an opportunity to iron out problems with the trial. If we find it is possible to run the trial on a small scale, we will apply for funding to run a full study. This will aim to answer the question of whether the continuous monitor improves the patient outcomes which were agreed during development with the patient public involvement group locally; rate of kidney damage, heart damage, stroke, post-operative infections, risk of death, and hospital length-of-stay.

Expected outcomes and implications. We anticipate we will find the trial to be feasible with amendments to the way it is run, and if this is the case, we will apply to run the full scale trial. If this shows that using the continuous monitor improves the patient outcomes above, then it would represent new, significant evidence that may lead to the NHS adopting it's use as 'standard care' during anaesthesia for repair of a broken hip, and would like lead to similar trials in other operations where patients may benefit in a similar way.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Adult patients, undergoing surgical repair of neck of femur fracture
3. Patient can understand and comprehend written and spoken English
4. Patient's consultee can understand written and spoken English

Exclusion Criteria:

1. American Society of Anaesthesiologists (ASA) Class I patients
2. Patients with device-specific exclusions; atrial fibrillation, Raynauds syndrome or disease, peripheral vascular disease, scleroderma, an arteriovenous shunt, valvular heart disease.
3. Patients in whom a blood pressure cuff cannot be safely inflated on both arms for any reason (for example, lymphoedema).
4. Patients in whom the treating anaesthetist has judged they will require invasive arterial pressure monitoring.
5. Patients declining consent
6. Patients in whom the treating anaesthetist will use total intravenous anaesthesia (TIVA)
7. Patients in whom there is a >20mmHg difference between non-invasive cuff mean arterial pressure measurements made on opposite arms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Feasibility Outcome - Proportion of recruited patients in whom CNAP was successfully applied and full data collected. | Through to study completion, an average of 5-6 weeks per patient.
  Proportion of recruited patients in whom CNAP was successfully applied and full data collected.
Feasibility Outcome - Proportion of eligible patients successfully recruited | Through to study completion, an average of 5-6 weeks per patient.
  The proportion of all those patients who are eligible during the recruitment period who are successfully enrolled into the trial.
Feasibility Outcome - Proportion of enrolled patients in whom there is a full data set recorded. | Through to study completion, an average of 5-6 weeks per patient.
Feasibility Outcome - Proportion of enrolled patients in which we are able to record full follow up data. | Through to study completion, an average of 5-6 weeks per patient.

SECONDARY OUTCOMES:
Intraoperative Outcomes - Nadir Blood Pressure | On the day of surgery only.
  The lowest mean arterial pressure recorded during surgery using the CNAP monitor
Intraoperative Outcomes - Total time spent with a mean arterial pressure <80mmHg | On the day of surgery only.
Intraoperative Outcomes - Total time spent with a mean arterial pressure <65mmHg | On the day of surgery only.
Intraoperative Outcomes - Total time spent with a mean arterial pressure <55mmHg | On the day of surgery only.
Intraoperative Outcomes - Total volume of intravenous fluids given | On the day of surgery only.
Intraoperative Outcomes - Total dose of vasopressors given | On the day of surgery only.
  Broken down into totals of each separate vasopressor used.
Post-operative Outcomes - Incidence of acute kidney injury in the 7 days post-operatively | Assessed up to 7 days post-operatively.
  Outcomes as per standardised definitions from the European Perioperative Clinical Outcome standards
Post-operative Outcomes - Incidence of myocardial injury in the first 3 days after surgery | Assessed up to 3 days post-operatively.
  Outcomes as per standardised definitions from the European Perioperative Clinical Outcome standards
Post-operative Outcomes - Incidence of stroke post-operatively | Assessed up to 30 days post-operatively.
  Outcomes as per standardised definitions from the European Perioperative Clinical Outcome standards
Post-operative Outcomes - Incidence of post-operative surgical site infection | Assessed up to 30 days post-operatively.
  As per CDC definitions
Post-operative Outcomes - Mortality | Assessed at 30 days post-operatively.
Health Economic Outcome - Hospital Length of Stay | Assessed at hospital discharge, an average of 10-14 days

CONTACTS AND LOCATIONS:
Locations (1):
- MIDRU, Birmingham Heartlands Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT04051073/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT04051073/ICF_001.pdf